CLINICAL TRIAL: NCT03183830
Title: A Double-blind, Randomised, Placebo-controlled Parallel Study to Investigate the Influence of Dietary Nitrate on Skin Inflammation in Healthy Volunteers
Brief Title: Influence of Dietary Nitrate on Skin Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16/LO/0160
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2018-06

CONDITIONS: Cardiovascular Diseases; Inflammation; Inflammation; Skin; Inflammatory Response; Nitric Oxide
Keywords: Cardiovascular Disease; Inorganic nitrate; Nitric Oxide; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation; Dermatitis

STUDY DESIGN:
Intervention Model Description: Double-blind randomised-control parallel two-limb study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All members of the study team and volunteer participants will be blinded to treatment versus placebo arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate-rich Beetroot Juice (Experimental): Individuals will receive a once daily dose of dietary nitrate in the form of a beetroot juice concentrate (70mL) containing ~5-6mmol inorganic nitrate (James White Drinks, UK) for 12 +/- 2 weeks. This dose has been chosen due to several reports demonstrating efficacy in patients with cardiovascular disease.
  Interventions: Dietary Supplement: Nitrate-rich Beetroot Juice
- Nitrate-deplete Beetroot Juice (Placebo Comparator): The placebo control is an identical juice from which the nitrate anion has been removed using a standard anion exchange resin. Visually there is no detectable difference between the juices and previous spectral, ion concentration, sugar levels, ascorbate analysis and taste testing has confirmed no differences in colour and constituents. The process to extract nitrate from the juice is the same technique used to remove inorganic nitrate from general drinking water supplies, and has been approved for use by Ethics Committees. The nitrate-free juice is not considered a drug or medicine, and is classified as a foodstuff.
  Interventions: Dietary Supplement: Nitrate-deplete Beetroot Juice

INTERVENTIONS:
Dietary Supplement: Nitrate-rich Beetroot Juice — The beetroot juice contains approximately 100kcal per 100mL of juice, equivalent to a glass of orange juice; the volume of juice per day for the study is 70mL. Volunteers will be informed that an average woman weighing 65kg should not consume more than 2000kcal per day, and an average man of 75kg not more than 2500kcal per day.
  Arms: Nitrate-rich Beetroot Juice
Dietary Supplement: Nitrate-deplete Beetroot Juice — See description of placebo juice in "Arms" for comparative information. The beetroot juice contains approximately 100kcal per 100mL of juice, equivalent to a glass of orange juice; the volume of juice per day for the study is 70mL. Volunteers will be informed that an average woman weighing 65kg should not consume more than 2000kcal per day, and an average man of 75kg not more than 2500kcal per day.
  Other Names: Placebo
  Arms: Nitrate-deplete Beetroot Juice

SUMMARY:
This study evaluates the potential anti-inflammatory effects of inorganic dietary nitrate in a model of acute inflammation relevant to cardiovascular disease (CVD).

Green leafy vegetables contain large amounts of inorganic nitrate, and research suggests that this nitrate has beneficial effects on the heart and blood vessels. The Ahluwalia Group have shown anti-inflammatory benefits of inorganic nitrate in pre-clinical models of CVD, early mechanistic studies in healthy volunteers, and in patients with hypertension, hypercholesterolaemia and those suffering acute heart attacks that translate to cardiovascular benefits. Understanding the mechanism of how this is achieved may open new therapeutic options in CVD.

The Investigators therefore wish to explore whether inorganic nitrate might alter inflammatory responses using a blister-model of acute skin inflammation. This study is a randomised control trial with parallel limbs where half of patients receive nitrate-rich beetroot juice, and the other half a nitrate-deplete placebo beetroot juice.

DETAILED DESCRIPTION:
Nitric oxide (NO) is an important substance produced continuously by all blood vessels. It is thought to maintain health, in part, by preventing and suppressing inflammatory responses. NO is normally generated at the endothelium by a group of important enzymes called nitric oxide synthases. However, in chronic inflammatory states such as those seen in cardiovascular disease (CVD), the endothelial isoform of the enzyme becomes dysfunctional and produces less NO, and the NO that is produced is scavenged by the products of oxidative stress.

Giving NO back to the blood vessel to mediate its beneficial effects is not straightforward. However, the Ahluwalia Group have shown that dietary inorganic nitrate, both as a capsule and a dietary intervention with nitrate-rich beetroot juice, has a number of beneficial effects in CVD states. This beneficial effect is mediated through it's endogenous conversion from nitrate to nitrite in the mouth, and then from nitrite to NO via nitrite reductases within the blood vessel. The Investigators have shown benefit of inorganic nitrate in pre-clinical models of CVD, early mechanistic studies in healthy volunteers, and anti-inflammatory benefits in patients with hypertension, hypercholesterolaemia and those suffering acute heart attacks.

The Investigators wish to prospectively investigate the anti-inflammatory effects of inorganic nitrate using a cantharidin-induced blister model of acute inflammation. This allows investigation of the innate immune system's response to an acute insult and characterise the inflammatory and resolution phases. Cantharidin is commonly used as a vesicant in the treatment of plantar verrucae and molluscum contagiosum, and experimentally to study the pharmacokinetics of drugs within the interstitial space.

This will be a double-blind placebo-controlled parallel limb study supplementing 24 healthy volunteers with dietary-rich beetroot juice versus nitrate-deplete placebo juice, to investigate blister formation, and inflammatory cell recruitment and activation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Caucasian
* Willing to provide informed consent

Exclusion Criteria:

* Healthy subjects unwilling to consent
* Non-caucasian volunteers
* History of any serious illnesses, including recent infections or trauma
* Subjects taking systemic medication (other than the oral contraceptive pill)
* Subjects with self-reported use of mouthwash or tongue scrapers
* Subjects with recent or current antibiotic use
* Subjects with a history, or recent treatment of (within last 3 months) any oral condition (excluding caries), including gingivitis, periodontitis and halitosis
* Subjects with a history of skin conditions
* Subjects with and history of allergic reaction to any topical application
* Subjects with any history of a bloodborne infectious disease such Hepatitis B or C virus, or HIV

We have excluded non-caucasian volunteers due to a small incidence of prolonged skin hyperpigmentation in non-caucasians in previous studies.

We have excluded subjects using mouthwash/tongue scrapers and oral conditions as we know that the nitrate ingested from the diet (i.e. beetroot juice) is converted to nitrite by the commensal bacteria in the back of the mouth. Subjects who have oral conditions or use mouthwash/tongue scrapers would have differences in oral bacterial populations, both in number and species. Therefore, by excluding these subjects, we will try and keep this variable as similar as possible in both groups.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change in plasma nitrate levels | 2 weeks
  Comparison of change in plasma nitrite following dietary nitrate or placebo supplementation
Change in blister fluid leucocytes | 2 weeks
  Comparison of change in blister fluid total and differential leucocyte numbers following dietary nitrate or placebo supplementation

SECONDARY OUTCOMES:
Change in blister fluid cytokine composition | 2 weeks
  Comparison of change in blister fluid cytokine analysis following dietary nitrate or placebo supplementation
Change in peripheral markers of inflammation | 2 weeks
  Comparison of change in peripheral markers of inflammation and leucocyte count following dietary nitrate or placebo supplementation
Change in non-invasive blood pressure measurement | 2 weeks
  Comparison of change in blood pressure following dietary nitrate or placebo supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Prof Amrita Ahluwalia, BSc PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
N/A - no plan to make IPD available to others

REFERENCES:
- [Background] Khambata RS, Ghosh SM, Rathod KS, Thevathasan T, Filomena F, Xiao Q, Ahluwalia A. Antiinflammatory actions of inorganic nitrate stabilize the atherosclerotic plaque. Proc Natl Acad Sci U S A. 2017 Jan 24;114(4):E550-E559. doi: 10.1073/pnas.1613063114. Epub 2017 Jan 5. PMID 28057862
- [Background] Rathod KS, Kapil V, Velmurugan S, Khambata RS, Siddique U, Khan S, Van Eijl S, Gee LC, Bansal J, Pitrola K, Shaw C, D'Acquisto F, Colas RA, Marelli-Berg F, Dalli J, Ahluwalia A. Accelerated resolution of inflammation underlies sex differences in inflammatory responses in humans. J Clin Invest. 2017 Jan 3;127(1):169-182. doi: 10.1172/JCI89429. Epub 2016 Nov 28. PMID 27893465
- [Background] Kapil V, Khambata RS, Robertson A, Caulfield MJ, Ahluwalia A. Dietary nitrate provides sustained blood pressure lowering in hypertensive patients: a randomized, phase 2, double-blind, placebo-controlled study. Hypertension. 2015 Feb;65(2):320-7. doi: 10.1161/HYPERTENSIONAHA.114.04675. Epub 2014 Nov 24. PMID 25421976
- [Background] Velmurugan S, Gan JM, Rathod KS, Khambata RS, Ghosh SM, Hartley A, Van Eijl S, Sagi-Kiss V, Chowdhury TA, Curtis M, Kuhnle GG, Wade WG, Ahluwalia A. Dietary nitrate improves vascular function in patients with hypercholesterolemia: a randomized, double-blind, placebo-controlled study. Am J Clin Nutr. 2016 Jan;103(1):25-38. doi: 10.3945/ajcn.115.116244. Epub 2015 Nov 25. PMID 26607938
- [Background] Jones DA, Pellaton C, Velmurugan S, Rathod KS, Andiapen M, Antoniou S, van Eijl S, Webb AJ, Westwood MA, Parmar MK, Mathur A, Ahluwalia A. Randomized phase 2 trial of intracoronary nitrite during acute myocardial infarction. Circ Res. 2015 Jan 30;116(3):437-47. doi: 10.1161/CIRCRESAHA.116.305082. Epub 2014 Dec 15. PMID 25512434
- [Background] Day RM, Harbord M, Forbes A, Segal AW. Cantharidin blisters: a technique for investigating leukocyte trafficking and cytokine production at sites of inflammation in humans. J Immunol Methods. 2001 Nov 1;257(1-2):213-20. doi: 10.1016/s0022-1759(01)00467-7. PMID 11687254
- [Derived] Lau C, Primus CP, Shabbir A, Chhetri I, Ono M, Masucci M, Bin Noorany Aubdool MA, Amarin J, Hamers AJ, Khan Z, Kumar NA, Montalvo Moreira SA, Nuredini G, Osman M, Whitear C, Godec T, Kapil V, Massimo G, Khambata RS, Rathod KS, Ahluwalia A. Accelerating inflammatory resolution in humans to improve endothelial function and vascular health: Targeting the non-canonical pathway for NO. Redox Biol. 2025 May;82:103592. doi: 10.1016/j.redox.2025.103592. Epub 2025 Mar 28. PMID 40209616